CLINICAL TRIAL: NCT02816099
Title: Study of the Influence of Glycaemic Balance on the Ability of Apolipoprotein C1 to Inhibit Cholesterol Ester Transfer Protein (CETP) in Type-1 Diabetes Patients
Brief Title: Influence of Glycaemic Balance on the Ability of Apolipoprotein C1 to Inhibit Cholesteryl Ester Transfer Protein in Type-1 Diabetes Patients
Acronym: ApoC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOUILLET AOI 2015
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: diabète de Type 1

ARMS (2):
- Type-1 diabetes patients (Experimental)
  Interventions: Biological: Prise de sang
- Controls (Other)
  Interventions: Biological: Prise de sang

INTERVENTIONS:
Biological: Prise de sang

SUMMARY:
In type-1 diabetes patients, bad cholesterol tends to accumulate because apoC1 function is slowed down.

ApoC1 is a protein whose role is to diminish the activity of CETP, another protein that regulates cholesterol transfer in the body.

The aim of this study is to determine whether it is possible to correct apoC1 function by improving glycaemic balance.

240 persons will be recruited in this study and allocated to one of two groups:

* 160 Type-1 diabetes patients with uncontrolled diabetes:

  * 4 additional blood samples will be taken at the time of the systematic biological examination at inclusion and then again 3 months later.
* 80 control subjects with normal lipids and normal glycaemia balance will be included in the study following the results of the biological assays.

  * 4 blood samples will be taken at the time of inclusion.

ELIGIBILITY:
Inclusion criteria for patients:

* Patients over 18 years
* Patients with type-1 diabetes and glycated hemoglobin (HbA1C) >9%

Inclusion criteria controls:

* Subjects over 18 years
* Normal glycaemia (Fasting glycaemia <1.10 g/L) and normal lipids (Low-density lipoproteins (LDL) <1.6 g/L, triglycerides (TG) <1.5 g/L)

Exclusion Criteria:

Exclusion criteria patients:

* Adults under guardianship
* Patients without national health insurance
* Pregnant or breast-feeding women
* Progressive cancer
* Treatment able to influence lipoprotein metabolism (oestroprogestatives, immunosuppressants, long-term corticotherapy)

Exclusion criteria controls:

* Adults under guardianship
* Persons without national health insurance
* Pregnant or breast-feeding women
* known dyslipidemia and/or lipid-lowering treatment
* Treatment able to influence lipoprotein metabolism (oestroprogestatives, immunosuppressants, long-term corticotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Comparaison of linear correlation coefficients between plasma concentrations of apoC1 and CETP activity | 3 mois

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besançon, Besançon
  - CHU Dijon Bourgogne, Dijon

REFERENCES:
- [Result] Rouland A, Gautier T, Denimal D, Duvillard L, Simoneau I, Rageot D, Verges B, Bouillet B. The Endogenous Inhibitor of CETP, apoC1, Remains Ineffective In Vivo after Correction of Hyperglycemia in People with Type 1 Diabetes. Metabolites. 2024 Sep 7;14(9):487. doi: 10.3390/metabo14090487. PMID 39330494
- [Derived] Denimal D, Monier S, Simoneau I, Duvillard L, Verges B, Bouillet B. HDL functionality in type 1 diabetes: enhancement of cholesterol efflux capacity in relationship with decreased HDL carbamylation after improvement of glycemic control. Cardiovasc Diabetol. 2022 Aug 12;21(1):154. doi: 10.1186/s12933-022-01591-9. PMID 35962339